CLINICAL TRIAL: NCT04018118
Title: Study of Clinical Profiles of Patients Followed for Chronic Hypereosinophilia and/or Hypereosinophilic Syndrome by the Creation of a National Cohort
Brief Title: Natural History of Hypereosinophilia and Hypereosinophilic Syndromes
Acronym: COHESION
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018_36; 2018-A02624-51 (Registry Identifier: ID-RCB - ANSM)
Record Dates: First submitted 2019-05-15; First posted 2019-07-12 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Eosinophilia; Hypereosinophilic Syndrome
Keywords: Eosinophilia; Hypereosinophilia; Hypereosinophilic Syndrome
MeSH Terms: conditions — Eosinophilia; Hypereosinophilic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Eosinophilia/Hypereosinophilic syndrome: patient with eosinophilia and/or hypereosinophilic syndrome
  Interventions: Biological: Biological sample

INTERVENTIONS:
Biological: Biological sample — Additional blood samples for biobanking

SUMMARY:
Unexplained chronic hypereosinophilia (HE) and hypereosinophilic syndromes (HES) are heterogeneous regarding the organ involvements (heart, lungs, skin, .. or none), the evolutionary profiles, the response to treatments.

Underlying mechanisms are largely unknown and may associate genetic predisposing factors (germinal ? somatic?), environmental factors (alimentation, tobacco use, hormones, infections, ..) The COHESion study aims to study all clinical and biological characteristics of HE/HES patients and their evolutionary profiles, with a focus on genetic factors and the mechanisms supporting transitory or persistant chronic HE/HES (in absence of any well identified extrinsic trigger like drugs, parasitosis, ..)

DETAILED DESCRIPTION:
There is currently no data on the natural history of unexplained chronic hypereosinophilia (HE) and hypereosinophilic syndromes (HES). Clinical practice shows that HE/SHE patients can present 4 evolutionary profiles:

A. a single flare-up of their disease, with favourable evolution spontaneously or under corticosteroid therapy, without further recurrence B. recurrent flare-ups with a variable free interval of several months to several years, with or without persistent eosinophilia between flare-ups C. a chronic disease requiring the continuation of a substantive treatment D. chronic asymptomatic HE for years: the mechanisms involved in the occurrence of possible organ damage are unknown

The primary objective of the study is to describe the frequency of the different clinical manifestations during the diagnostic and follow-up of the hypereosinophilic syndrome (HES). The primary endpoint is the frequency of the different clinical manifestations and/or organs damage related to eosinophilia.

ELIGIBILITY:
Inclusion Criteria:

* Men or Women of any age :
* With the diagnosis criteria of hyperosinophlia OR hypereosinophilic syndrome OR specific organ eosinophilic disease according to the consensus conference of the International Cooperative Working Group on Eosinophil Disorders (ICOG-EO)
* With an AEC > 1500/mm3 or organ damage related to the presence of eosinophils in the tissues or organs whatever the context (idiopathic, clonal or reactive, including drug-related, parasitic or allergic)
* HES diagnosis since 2005/01/01
* Patients socially insured
* Patient who agreed to participate to the study, its proceedings and duration.

Exclusion Criteria:

* Known HIV infection
* Not socially insured
* Person unable to receive a enlighten information
* Person who refuse to sign the consent
* Persons deprived of their liberty
* Persons benefiting from a system of legal protection (tutelage / guardianship)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Hypereosinophilia and Hypereosinophilic Syndromes
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-05-06 (Actual); Primary Completion 2029-05-06 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
Frequency of the different clinical manifestations at time of diagnosis and during follow-up of the hypereosinophilic syndrome (HES) | 10 years
  The primary objective of the study is to describe the frequency of the different clinical manifestations at diagnosis and during follow-up of the hypereosinophilic syndrome (HES/HE). The primary endpoint is the frequency of the different clinical manifestations and/or organs damage related to hypereosinophilia.

SECONDARY OUTCOMES:
Frequency of the evolutionary profiles | 10 years
  Frequency of the different evolutionary profiles.
Frequency of complications depending of the type of HES | 10 years
  Frequency of complications (organ damages) depending on the type of HES (idiopathic, reactive, clonal…).
Frequency of organ damage profiles before and after 18 years old. | 10 years
  Describe the characteristics of pediatrics HE/HES vs adult HE/HES.
Frequency of clinical complications profiles before and after 18 years old. | 10 years
  Clinical characteristics of pediatrics HE/HES vs adult HE/HES.
Frequency of HLA alleles and variants / mutations on other genes of HE/HES | 10 years
  Predisposing factors in HE/HES by various genomic approaches
Serum biomarkers | 10 years
  to explore Potential predisposing factors in HE/HES: serum markers predictive of interest in eosinophilopoiesis (IL5), tissue homing (eotaxins, etc.)
Difference in Membrane activation markers of HE patients (asymptomatic) versus SHE (symptomatic). | 10 years
  Predisposing factors in HE/HES by various genomic approaches
Difference in Eosinophilic gene expression profiles of HE patients (asymptomatic) versus SHE (symptomatic). | 10 years
  Predisposing factors in HE/HES by various genomic approaches

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Lefevre, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHU, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lefevre G, Bleuse S, Puyade M, Moulis G, Neel A, Abisror N, Baudet A, Bonnotte B, Dion J, Dossier A, Grall M, Lifermann F, Limal N, Lioger B, Machelart I, Mohr C, Outh R, Queyrel-Moranne V, Slama B, Trefond L, Abou Chahla W, Ackerman F, Belfeki N, Berezne A, Blade JS, Bouderbala MA, Chebrek S, Cottin V, De Almeida S, De Masson A, Dezoteux F, Goulenok T, Jachiet V, Jouvray M, Latu I, Ledoult E, Leurs A, Lugosi M, Martin M, Melboucy-Belkhir S, Morati-Hafsaoui C, Quemeneur T, Rohmer J, Roy-Peaud F, Sanges S, Schleinitz N, Staumont-Salle D, Taille C, Terriou L, Tieulie N, Koenga JDE, Schwarb L, Panel K, Kahn JE, Groh M; COHESion study group. Hypereosinophilia and Hypereosinophilic Syndromes: First Findings From a Nationwide Multicenter Cohort. Allergy. 2025 Apr;80(4):1100-1110. doi: 10.1111/all.16463. Epub 2025 Jan 5. PMID 39757773